CLINICAL TRIAL: NCT06672913
Title: Impact of Standardized Skin-to-Skin Care on Clinical Outcomes in Infants Born ≤ 32 Weeks: A Multicenter Study
Acronym: TR-SSCinNICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Collaborators: Ankara University (Other); Gazi University (Other); Hacettepe University (Other); Marmara University (Other); Umraniye Education and Research Hospital (Other Government); Trakya University (Other); Ege University (Other); Ondokuz Mayıs University (Other); Cukurova University (Other); Sanliurfa Harran University (Unknown); Cumhuriyet University (Other); Uludag University (Other); Kocaeli University (Other); Aydin Adnan Menderes University (Other); Konya City Hospital (Other); Baskent University (Other)
Responsible Party: Principal Investigator, Sezin Unal, Prof, MD, Baskent University Ankara Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TR-SSCinNICU
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Premature; Skin to Skin Contact; Breast Feeding; Necrotizing Enterocolitis; Retinopathy of Prematurity
Keywords: Premature; Skin to skin contact; Breast Feeding; Necrotizing Enterocolitis; Retinopathy of Prematurity
MeSH Terms: conditions — Premature Birth; Breast Feeding; Enterocolitis, Necrotizing; Retinopathy of Prematurity

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective pre and post training interventional clinical study. The effect of a standardized skin-to-skin contact application, which is initiated early and applied regularly, on clinical outcomes for preterm infants born at less than 32 weeks of gestation will be investigated.
  Intervention: Teoritical and practical education on skin to skin contact to ensure the application of Turkish Neonatal Society skin to skin contact protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre education (No Intervention): The infants born at less than 32 weeks and discharged from the units in the last two months before training.
- Post education (Active Comparator): The infants born at less than 32 weeks and discharged between four to six months after training
  Interventions: Behavioral: skin to skin contact care

INTERVENTIONS:
Behavioral: skin to skin contact care — Early and regular skin to skin contact in NICU GA: < 28 weeks: After the 72nd hour GA: 28 - 32 weeks: As soon as stabilization is ensured
  Arms: Post education

SUMMARY:
This study is a multi-center, prospective pre-post clinical study conducted under the leadership of the Turkish Neonatal Society. It aims to investigate the effects of a standardized skin-to-skin care in NICU, initiated early and applied regularly, on recieving exclusive mothers' milk at discharge and clinical outcomes for preterm infants born ≤ 32 weeks of gestation.

1. Primary Objective: To evaluate the rate of receiving exclusive mothers' milk at discharge for infants born ≤ 32 weeks of gestation who have received skin-to-skin care in accordance with the study protocol.
2. Secondary Objective: To evaluate the rates of neonatal sepsis, intraventricular hemorrhage, and necrotizing enterocolitis (stage 2 and above) as well as the length of hospital stay for infants born at or below 32 weeks of gestation who have received skin-to-skin care in accordance with the study protocol.

DETAILED DESCRIPTION:
1. Introduction: Throughout the historical evolution of the field of neonatology, negative consequences of newborns being separated from their families for extended periods while in neonatal intensive care units (NICUs) have been observed. In 1978, the concept of "Skin-to-skin care: Kangaroo Mother Care" was introduced. This model has been recommended by the World Health Organization to replace incubators and radiant warmer technologies in developing and least developed countries, where the capacity of NICUs is very limited. Additionally, in developed countries, where newborn health indicators are optimal, family-centered care and family-integrated care approaches have been used as crucial components to maintain the bond between mothers-and even families-with patients requiring NICU care and premature newborns. Canada in North America and Scandinavian countries in Europe are pioneers of this approach. In developed countries that have adopted this model, regardless of how small, premature, or ill the newborn is, their medical needs are met from birth while ensuring skin-to-skin care with their mother or father. In today's changing architecture of NICUs, care and treatment are conducted in "personalized neonatal intensive care areas for families," with the participation of families.

   Skin-to-skin care has been shown to be effective in improving breastfeeding rates, enhancing bonding, better physiological stability, reducing stress levels, shortening hospital stays, decreasing the risk of infections, lowering rates of intraventricular hemorrhage, and improving weight gain and parental confidence. Additionally, it has been shown to be most effective when skin-to-skin care is applied for more than one hour in a single session and for more than eight hours in a day. This can be best assured if a protocol exists in the units.
2. Objective: This study is a multi-center, prospective pre-post clinical study conducted under the leadership of the Turkish Neonatal Society. It aims to investigate the effects of a standardized skin-to-skin care application, which is initiated early and applied regularly, on clinical outcomes for preterm infants born at less than 32 weeks of gestation.

   1. Primary Objective: To evaluate the rate of receiving exclusive mothers' milk at discharge for infants born ≤ 32 weeks of gestation who have received skin-to-skin care in accordance with the study protocol.
   2. Secondary Objective: To evaluate the rates of neonatal sepsis, intraventricular hemorrhage, and necrotizing enterocolitis (stage 2 and above) as well as the length of hospital stay for infants born at or below 32 weeks of gestation who have received skin-to-skin care in accordance with the study protocol.
3. Method: Eight training institutions (hospitals) from different geographical regions of Turkiye will be selected. Once the chair of the selected NICUs express their consent to participate, detailed information about the project will be provided to them. The training program developed regarding the skin-to-skin care approach will be delivered in a face-to-face format on a full training day for the responsible physicians and nursing staff working in the units. The theoretical lesson program will consist of three 45-minute lessons (history, standard skin-to-skin care application, skin-to-skin care application for at-risk infants). Practical lessons will be conducted in pairs using a realistic scenario with models. Following the theoretical and practical lessons, the aim is to implement skin-to-skin care based on a standardized protocol for at least one hour per each session, initiated early and regularly.

   a. The skin-to-skin care application proposed by the Turkish Neonatology Association is as follows:

   i. Duration: At least one hour per session

   ii. Time to initiate first skin-to-skin care:

   GA: < 28 weeks: After the 72nd hour GA: 28 - 32 weeks: As soon as stabilization is ensured

   iii. Criteria to accepted as stabilization: Absence of hypothermia Normal arterial tension with or without inotropic treatment Vital signs stable or easily normalized after nursing care Absence of frequent (>3/hour) and profound (any apnea requiring positive pressure ventilation in the last three hours) apnea

   b. Data Recording: Feeding details at discharge (Exclusive mothers'milk, ≥ 50% mothers' milk, < 50% mothers' milk, Formula) and data regarding outcomes (sepsis, intraventricular hemorrhage, necrotizing enterocolitis, duration of hospitalization) will be recorded for patients in the pre-education and post-education groups in each unit. The pre-education group includes infants discharged from the units in the two months prior to training, while the post-education group includes infants discharged from the units between the fourth and sixth months after training. Data collected before and after the intervention will be analyzed.

   c. Sample Size: To determine the sample size, a power analysis was conducted using the OpenEpi program. Assuming a 95% confidence level (1-α), an 80% test power (1-β), and an expected effect size of d=0.25, it was determined that at least 59 samples are required in each group.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at gestational age ≤ 32 weeks

Exclusion Criteria:

* Death before NICU discharge
* Abdominal wall defects

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Mothers' Milk at Discharge | Through study completion, an average of 3 months, at the time of discharge
  Number of infants receiving Exclusive Mothers' Milk at Discharge

SECONDARY OUTCOMES:
Intraventricular hemorrhage | Through study completion, an average of 3 months, at the time of discharge
  Number of infants with intraventricular hemorrhage diagnosed by cranial ultrasound
Necrotizing enterocolitis (stage 2 and above) | Through study completion, an average of 3 months, at the time of discharge
  Number of infants with necrotizing enterocolitis (stage 2 and above) according to Bell's criteria
Early neonatal sepsis | Through study completion, an average of 3 months, at the time of discharge
  Number of infants with sepsis within first three days of admission; culture positive or clinical
Late neonatal sepsis | Through study completion, an average of 3 months, at the time of discharge
  Number of infants with sepsis after the third day of admission; culture positive or clinical
Length of hospital stay | Through study completion, an average of 3 months, at the time of discharge
  Total length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Esin Koc, Prof, MD, Study Chair — Gazi University; Saadet Arsan, Prof, MD, Study Director — Ankara University; Hülya Bilgen, Prof, MD, Study Director — Marmara University; İlke Mungan Akın, Prof, MD, Study Director — Umraniye Teaching and Research Hospital; Betül Acunaş, Prof, MD, Study Director — Trakya University; Mehmet Yalaz, Prof, MD, Study Director — Ege University; Sezin Unal, Prof, MD, Study Director — Baskent University; Sule Yigit, Prof, MD, Study Director — Hacettepe University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No